CLINICAL TRIAL: NCT06077370
Title: Effectiveness of Deep Transcranial Magnetic Stimulation to Medial Prefrontal Cortex and Anterior Cingulate Cortex in Obsessive-Compulsive Disorder Patients
Brief Title: dTMS in Obsessive Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Selim Tumkaya, Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021TIPF029
Record Dates: First submitted 2023-09-27; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: obsessive compulsive disorder; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dTMS group (Active Comparator): dTMS on anterior cingulate cortex and medial prefrontal cortex.
  Interventions: Device: deep TMS
- sham TMS (Sham Comparator): Sham TMS on anterior cingulate cortex and medial prefrontal cortex.
  Interventions: Device: Sham TMS

INTERVENTIONS:
Device: deep TMS — Deep Transcranial magnetic stimulation on anterior Cingulate cortex and medial prefrontal cortex. 20 Hz.
  Arms: dTMS group
Device: Sham TMS — Sham Transcranial magnetic stimulation on anterior Cingulate cortex and medial prefrontal cortex. 20 Hz.
  Arms: sham TMS

SUMMARY:
High-frequency deep transcranial magnetic stimulation (dTMS) over the medial prefrontal cortex (mPFC) and the anterior cingulate cortex (ACC) with an H-coil has been approved by the Food and Drug Administration for use in treatment-resistant obsessive-compulsive disorder (OCD). However, there is not yet strong scientific evidence concerning the efficacy and safety of performing a similar procedure with a double-cone coil or in an accelerated manner. The aim of this study was evaluating the efficacy of dTMS over the medial prefrontal cortex (mPFC) and the anterior cingulate cortex (ACC) in an accelerated manner with double-cone coil.

DETAILED DESCRIPTION:
The current study aimed to investigate the efficacy and safety of multiple deep stimulations per day with a double-cone coil to the mPFC and ACC in treatment-resistant patients with OCD. This study evaluated (I) the effectiveness of high-frequency stimulation of the mPFC and ACC with a double cone coil, and (II) the effectiveness of the application of this protocol in three weeks, not six weeks as approved by the FDA. The participants were randomized into two parallel groups in a double-blind manner. High frequency (20 Hz) dTMS was applied to the mPFC and ACC in one group and sham dTMS to the same regions in the other group, twice a day, for a total of 30 sessions. This application was for three weeks in total, excluding weekends.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of obsessive-compulsive disorder
* Not having an adequate response to treatment despite using at least two selective serotonin reuptake inhibitors at a sufficient dose and duration for 12 weeks before the planned add-on treatment
* Aged 18-65 years
* Able to read and write

Exclusion Criteria:

* Not providing consent to participate in the study
* Diagnosis of a psychiatric disorder, such as psychotic disorder, bipolar disorder, major depressive disorder [Hamilton Depression Rating Scale (HDRS) score above 17], mental retardation, alcohol-substance use disorder, and organic mental disorder (dementia, delirium, and head trauma, etc.)
* Diagnosis of an important medical or neurological disease (e.g., epilepsy);
* Mental retardation
* Illiteracy
* Having received electroconvulsive therapy (ECT) or TMS within the last six months;
* Having any prosthesis, such as an implant and pacemaker.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-11-27 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Obsessive compulsive symptoms severity | pretreatment(0.weeks)-as soon as the work is completed (3 weeks)
  Yale-Brown Obsessive-Compulsive Scale (Y-BOCS). The minimum and maximum values are 0-40, and higher scores mean a worse outcome.
Dimensional obsessive compulsive symptom severity | pretreatment(0.weeks)-as soon as the work is completed (3 weeks)
  Dimensional Obsessive-Compulsive Scale (DOCS). The minimum and maximum values are 0-80, and higher scores mean a worse outcome.
Severity of side effects | pretreatment(0.weeks)-as soon as the work is completed (3 weeks)
  Clinical Global Impression - The efficacy index. The minimum and maximum values are 1-4, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Severity of Depression | pretreatment(0.weeks)-as soon as the work is completed (3 weeks)
  Hamilton Depression Rating Scale. The minimum and maximum values are 0-52, and higher scores mean a worse outcome.
Severity of anxiety | pretreatment(0.weeks)-as soon as the work is completed (3 weeks)
  Hamilton Anxiety Rating Scale. The minimum and maximum values are 0-56, and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Selim Tümkaya, MD, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No